CLINICAL TRIAL: NCT02939443
Title: Diagnosis of Inguinal Hernia by Prone- vs. Supine-position Computed Tomography
Brief Title: Prone-position CT for Diagnosing Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagareyama Central Hospital (Other)
Responsible Party: Principal Investigator, Akira Miyaki, chief of surgery department, Nagareyama Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCH 14-3
Record Dates: First submitted 2016-10-14; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Supine Position

ARMS (1):
- cross-sectional study (Other)
  Interventions: Radiation: supine- and prone-position Computed Tomography

INTERVENTIONS:
Radiation: supine- and prone-position Computed Tomography

SUMMARY:
Background: The aim of this study was to investigate the efficacy of prone-position computed tomography (CT) for detecting and classifying inguinal hernia relative to supine-position CT before laparoscopic inguinal hernia repair.

Materials and Methods: Sixty-eight patients who underwent laparoscopic transabdominal preperitoneal repair of inguinal hernia were enrolled in this prospective study. Patients diagnosed with inguinal hernia by physical examination underwent abdominal CT in the supine and prone positions for preoperative assessment. The anatomy of the right and left inguinal regions was confirmed during the surgery and compared with the preoperative CT findings.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia

Exclusion Criteria:

* emergency surgery for incarcerated hernia
* femoral hernia
* recurrent inguinal hernia after laparoscopic inguinal hernia repair

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The detection rate of inguinal hernia | two years